CLINICAL TRIAL: NCT04199182
Title: Exploring the Effects of Exercise Training on PTSD Symptoms and Physical Health in Older Veterans With PTSD
Brief Title: Exercise Training to Improve PTSD Symptoms and Health in Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3120-R; RX003120 (Other Grant/Funding Number: VAORD)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Physical performance; Veterans; Aged; Exercise; HRQOL
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Behavioral intervention testing the effects of supervised exercise versus attention-control on PTSD symptoms and function.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Progressive, multi-component supervised exercise training group.
  Interventions: Behavioral: Exercise Training
- Healthy Aging Attention Control (Active Comparator): A health education program that addresses topics relevant to older adults.
  Interventions: Other: Healthy Aging Attention Control (HA-ATC)

INTERVENTIONS:
Behavioral: Exercise Training — A multi-component group exercise intervention that emphasizes functional training. Duration is 6 months, and frequency is 3x per week.
  Arms: Exercise
Other: Healthy Aging Attention Control (HA-ATC) — Participants in the HA-ATC group will receive a health education program modeled on the "10 Keys to Healthy Aging" curriculum and the National Council on Aging's "Aging Mastery Program." HA-ATC will include an 8-week face-to-face group program followed by bi-weekly sessions for the remaining 4 months.
  Other Names: HA-ATC
  Arms: Healthy Aging Attention Control

SUMMARY:
Posttraumatic stress disorder (PTSD) is prevalent among military Veterans and is more than just a psychological condition; PTSD has profound negative impacts on health, function, and quality of life. Older Veterans are the largest patient population served by the Veterans Health Administration (VHA), and many have lived with PTSD for 40+ years. Veterans with PTSD engage in low levels of physical activity and spend much of their time in sedentary activities, adding to their risk of physical disability. The benefits of exercise on mental health and physical well-being in older adults are well-substantiated, but the effects of exercise training on late-life PTSD symptoms is a new area of study. This study is designed to examine the effects of 6 months of supervised exercise training on PTSD symptoms and PTSD-related conditions (e.g., functional impairment, sleep) in 188 older Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* registered for care at Durham VA Health Care System (VAHCS)
* live within 50 miles of fitness facility
* meet diagnostic criteria for PTSD as assessed by the CAPS-5

Exclusion Criteria:

* history of any psychiatric disorder with severe psychotic features in the past 5 years (e.g., bipolar disorder, mania), as indicated by ICD-10 codes F20-F29 (ICD-9 category 298.9)
* prominent suicidal ideation or hospitalization for suicidality in the previous 6 months
* clinically significant: neurological disorder, systemic illness affecting central nervous system (CNS) function, or history of seizure disorder in the past 5 years
* uncontrolled diabetes defined as:

  * Abnormal fasting plasma glucose 126 mg/dL, random plasma glucose 200 mg/dL
  * no active medications for diabetes management (Metformin, insulin, etc.)
  * no clinical notes in the patient's electronic health record (EHR) indicating monitoring by primary care physician (PCP) or Endo for diabetes management)
  * end stage liver disease or currently receiving dialysis
  * physical disabilities precluding use of exercise equipment (assistive mobility devices acceptable)
  * significant cognitive impairment or diagnosis of Alzheimer's Disease or Dementia
  * hospitalization or ER visit in the past 6 months for conditions contraindicated for exercise (cardiac event; physical trauma)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-V (CAPS-5) | 6 months
  PTSD symptoms over the previous month will be assessed with the CAPS-5 clinical interview. Total symptom severity score and symptom cluster severity scores will be calculated. Scores range from 0 to 80, with higher scores reflecting more sever PTSD symptoms.
Six-minute walk test | 6 months
  Performance-based measure of aerobic endurance. Participants are instructed to walk along a measured course for 6 minutes. The distance walked in 6 minutes (feet) is the outcome of this assessment. There is no maximum value for this test, but the minimum value could be 0 (unable to walk any distance).

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 6 months
  Self-report tool for assessing the severity of depression. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Pittsburgh Sleep Quality Index (PSQI) | 6 months
  The PSQI is a self-report tool for assessing sleep quality and disturbance. Scores on the PSQI range from 0 to 21, with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Shepherd Hall, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification, will be made available.
  A limited dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Only de-identified (stripped of 18 HIPAA) and anonymized datasets (void of any identifying code, study or otherwise) will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available immediately following publication. No end date.
Access Criteria: Requests for de-identified meta-data will be considered by the PI, under a data-sharing agreement that includes: 1) a commitment to using the data only for research purposes; 2) a commitment to securing data using appropriate digital technology; and 3) a commitment to destroying or returning the data after analyses are complete. Data access will be provided only to qualified researchers, with a methodologically sound proposal, fully consistent with the VA/NIH data sharing policies and applicable laws and regulations.

DOCUMENTS (1):
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT04199182/ICF_000.pdf